CLINICAL TRIAL: NCT02705209
Title: Cayenne Pepper Cataplasm - Effect Study on Healthy Subjects and Subjects With Back Pain
Brief Title: Cayenne Pepper Cataplasm - Effect Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation (Other)
Collaborators: Comenius University (Other)
Responsible Party: Principal Investigator, Helmut Kern, MD PhD, Univ.-Prof. DDr., Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Munari02
Record Dates: First submitted 2015-10-23; First posted 2016-03-10 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Back Pain; Low Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Other: Cayenne Pepper Cataplasm
- Control (Placebo Comparator)
  Interventions: Other: Placebo Cataplasm

INTERVENTIONS:
Other: Cayenne Pepper Cataplasm — Poultice of Kaolin, Cayenne Peppfer (5%) and Water
  Arms: Treatment
Other: Placebo Cataplasm — Poultice of Kaolin and Water
  Arms: Control

SUMMARY:
The beneficial analgesic effects of Rubefacenciae (redden skin substances), is known since 1830 as a treatment for pain, cramps, and disorders of the musculoskeletal system. Herbal cataplasms containing rubefacient substances, such as Cayenne pepper, are commonly used as natural medications to treat painful or aching areas in the case of acute or chronic back pain, and rheumatisms. In Vienna and lower Austria, a Cayenne Pepper Cataplasm (CPC) application containing Cayenne pepper and Kaolin powder in mixed proportion, is commonly used to treat musculoskeletal conditions of pain especially of the low back.

Therefore, the aim of the present study was to test effects of a series of ten applications of CPC prepared with 5% of pepper, investigating the resulting effect on: skin temperature, skin sensory functions, pain threshold, and proprioception. Placebo control condition (0% cayenne pepper) was also tested. It was hypothesized that a series of 20-minute application of a CPC will have significant effects on the measured parameters.

40 subjects will be randomized into Treatment/control group.

ELIGIBILITY:
Inclusion Criteria:

* chronic lumbar spine pain >= 3 months
* pain during activity VAS >= 4
* Oswestry Disabilty Index >= 20%

Exclusion Criteria:

* pregnancy
* sensibility disorders (e.g. due to neurological disease)
* injuries, open wounds or rash in intervention area
* known hypersensitivity against the applied substances
* HIV, Hepatitis C and other due blood communicable infectious diseases

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Two-point discrimination test | before 1st and 3 weeks later after 10th intervention
  The subject is lying prone during the test and test will be performed with a BASELINE Aesthesiometer (0-100mm). The test will be performed at the level of L3 spinal process, the medial pin 3 cm laterally from midline and the pins oriented in medial-lateral direction. The two pins will be pressed perpendicular to the skin and the subject will be asked to report whether he/she feels one or two pins. Each inter-pin distance will be used three times using single pin touches in between for a control. The smallest inter-pin distance which the subject reports correctly at least 2 out of 3 repetitions, will be taken, as the result of the test.

SECONDARY OUTCOMES:
Monofilament Test | before 1st and 3 weeks later after 10th intervention
  Different monofilaments (Semmes-Weinstein) will be randomly pressed perpendicular to the same area as primary outcome measure. The thinest filament recognized from the subject will be taken as the result of the test.
Skin Temperature | before 1st and 3 weeks later after 10th intervention
  measured via Infrared thermometer
Blood Sample | before, 1h and 48h after the first intervention and 3 weeks later before, 1h and 48h after 10 interventions
  test: hemogram, CRP, CK, blood sedimentation rate, albumin and different molecular markers
Range of Motion (thoracic and lumbar spine) | before 1st and 3 weeks later after 10th intervention
  Measured according to Schober and Ott test

CONTACTS AND LOCATIONS:
Locations (2):
- Ludwig Boltzmann Institute of Electrical Stimulation and Physical Rehabilitation, Vienna, Austria
- Facultiy of Physical Education and Sports, Comenius University of Bratislava, Bratislava, Slovakia